CLINICAL TRIAL: NCT00111514
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalating Study to Evaluate Safety, Tolerability, and Immunogenicity of Leish-111f + MPL-SE Vaccine in Combination With Pentavalent Antimony in Treatment of Mucosal Leishmaniasis
Brief Title: Study to Evaluate the Leish-111F + MPL-SE Vaccine in the Treatment of Mucosal Leishmaniasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDRI-LMVTC-102
Record Dates: First submitted 2005-05-20; First posted 2005-05-23 (Estimated); Last update posted 2007-02-15 (Estimated); Status verified 2007-02

CONDITIONS: Leishmaniasis, Mucocutaneous
Keywords: Leishmaniasis; Subunit vaccine; therapeutic; T-cell; pentavalent antimony
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous; Leishmaniasis

INTERVENTIONS:
Biological: Leish-111f + MPL-SE vaccine

SUMMARY:
The purpose of this study is to evaluate the safety of the Leish-111f + MPL-SE vaccine given as three injections every 28 days at each of three dose levels of Leish-111f protein, in combination with standard pentavalent antimony therapy in adult patients with mucosal leishmaniasis.

DETAILED DESCRIPTION:
Mucosal leishmaniasis is a disfiguring and possibly fatal infection. All available medical therapies require weeks of treatment and cause significant toxicity. In Peru, the standard therapy is daily intravenous (IV) pentavalent antimony (20 mg/kg/day) for 28 days. It appears that Leishmania infections can be eliminated by T helper 1 immune responses. These findings argue that a vaccine that augments mucosal leishmaniasis patients' T helper 1 responses will eliminate the infection and disease. This study is a phase 1, randomized, double-blind, placebo controlled, sequential dose-escalating trial to evaluate the safety and immunogenicity of three injections of 5, 10, or 20 μg of Leish-111f protein + 25 μg of MPL-SE adjuvant given at 4 week intervals as an adjunct to standard chemotherapy with pentavalent antimony (20 mg/kg/day for 28 days) in patients with mucosal leishmaniasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mucosal leishmaniasis confirmed by a positive smear, in vitro culture or PCR test

Exclusion Criteria:

* Mucosal leishmaniasis must not involve the vocal cords or cause respiratory distress, and there must be no evidence of other disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48
Dates: Start 2004-07; Study Completion 2006-05

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicity
Adverse events

SECONDARY OUTCOMES:
IgG and T-cell response to Leish-111f vaccine
Leish-111f skin test reactivity
Safety of the vaccine with respect to the clinical course of mucosal leishmaniasis

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Llanos-Cuentas, MD, Principal Investigator — Universidad Peruana Cayetano Heredia; Franco M Piazza, MD, MPh, Study Director — Access to Advanced Health Institute (AAHI)
Locations (2):
- Peru (2):
  - Clínica de Leishmaniasis, Hospital Nacional Sur Este EsSalud, Cusco
  - Universidad Peruana Cayetano Heredia, Lima

REFERENCES:
- [Derived] Llanos-Cuentas A, Calderon W, Cruz M, Ashman JA, Alves FP, Coler RN, Bogatzki LY, Bertholet S, Laughlin EM, Kahn SJ, Beckmann AM, Cowgill KD, Reed SG, Piazza FM. A clinical trial to evaluate the safety and immunogenicity of the LEISH-F1+MPL-SE vaccine when used in combination with sodium stibogluconate for the treatment of mucosal leishmaniasis. Vaccine. 2010 Oct 28;28(46):7427-35. doi: 10.1016/j.vaccine.2010.08.092. Epub 2010 Sep 17. PMID 20851080